CLINICAL TRIAL: NCT03771352
Title: A Prospective Multi-Center Clinical Study to Evaluate Uncorrected Distance Vision and Quality of Vision After Light Treatments of an Implanted RxSight Light Adjustable Lens (RxLAL) With the Light Delivery Device (LDD) in Subjects With Preoperative Corneal Astigmatism
Brief Title: Clinical Study to Evaluate the RxSight Light Adjustable Lens With the Light Delivery Device in Subjects With Preoperative Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-025-03
Record Dates: First submitted 2018-11-30; First posted 2018-12-11 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Cataract
Keywords: cataract surgery; eye disease; lenticular opacification
MeSH Terms: conditions — Cataract; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- RxSight RxLAL IOL (Other): Eligible patients will be implanted with the RxSight RxLAL intraocular lens (IOL)
  Interventions: Device: RxSight RxLAL

INTERVENTIONS:
Device: RxSight RxLAL — The patients will be assessed for 6 months
  Other Names: Light Adjustable Lens; Light Delivery Device

SUMMARY:
For patients undergoing cataract surgery, the purpose of this study is to evaluate a patient's far vision without glasses and quality of vision after implantation and UV treatment of the RxSight Light Adjustable Lens (RxLAL).Following completion of all light treatments, the patient's far vision without glasses and quality of vision will be assessed 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Must sign a written Informed Consent form and be willing to undergo cataract surgery for the bilateral implantation of the RxLAL.
* Greater than the age of 40 on the day the cataract surgery is performed.
* Preoperative keratometric cylinder of >=0.50 D and <=4.00 D in both eyes.
* Cataract causing reduction in best corrected distance visual acuity (BCDVA) to a level of 20/32 or worse with or without glare source in both eyes.
* Willing and able to comply with the requirements for study specific procedures and visits.

Exclusion Criteria:

* Zonular laxity or dehiscence.
* Age-related macular degeneration involving the presence of geographic atrophy or soft drusen.
* Retinal degenerative disorder or macular disorder (other than mild macular degeneration) that is expected to cause future vision loss.
* History of uveitis
* Keratoconus or suspected of having keratoconus.
* Previous corneal or intraocular surgery, except eyes with previous pterygium excision are permitted as long as the pterygium did not extend more than 2mm onto the cornea from the limbus.
* Serious co-morbid conditions that in the judgement of the investigator makes inclusion in the study not in the best interest of the subject.
* Subjects taking systemic medications that may increase sensitivity to UV light.
* Subjects taking a systemic medication that is considered toxic to the retina such as tamoxifen.
* History of ocular herpes simplex virus
* History of congenital color vision defect

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Dick, MD, Principal Investigator — University Eye Clinic- Bochum, Germany; Fritz Hengerer, MD, Principal Investigator — University Eye Clinic- Heidelberg, Germany; Sathish Srinivasan, MD, Principal Investigator — Ayrshire Eye Clinic and Laser Center
Locations (3):
- Germany (2):
  - University Eye Clinic, Bochum
  - University Eye Clinic, Heidelberg
- Ayrshire Eye Clinic and Laser Center, Ayr, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | RxSight RxLAL IOL
Started | 55; 110 Eyes
Completed | 51; 101 Eyes (The fellow eye of one subject was not implanted per the discretion of the investigator.)
Not Completed | 4; 9 Eyes
Not completed — Screen failure | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | RxSight RxLAL IOL
Number analyzed (Participants) | 51
Number analyzed (Eyes) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0
  Black or African American | 0
  White | 51
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8
  Germany | 43
Primary Eyes Enrolled [Count of Units; unit: Eyes] — Subjects dominant eyes were assigned to the Primary Eye Enrolled group. Population: "Primary eyes enrolled" represent a count of units distributed across mutually exclusive and exhaustive categories
  Eyes
    number analyzed (Eyes) | 51
    OD | 26
    OS | 25
Fellow Eyes Enrolled [Count of Units; unit: Eyes] — Subjects non- dominant eyes were assigned to the Fellow Eye Enrolled group. Population: "Fellow eyes enrolled" represent a count of units distributed across mutually exclusive and exhaustive categories
  Eyes
    number analyzed (Eyes) | 50
    OD | 24
    OS | 26

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Distance Visual Acuity (UCDVA) of 20/20 or Better
Description: Percent of eyes with monocular uncorrected distance visual acuity of 20/20 or better
Time Frame: at 6 months postop
Population: A modified Effectiveness (m-Effectiveness) population was used for all effectiveness analyses which includes all observed data without treatment related protocol deviations.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | RxSight RxLAL IOL
Number analyzed (Participants) | 30
Number analyzed (Eyes) | 59
Eyes | 45

2. Other Pre Specified Outcome: Safety: ISO 11979-7 Ocular Adverse Events (Device Related and Unrelated)
Description: Number of study eyes experiencing Ocular adverse events (device related and unrelated)
Time Frame: Through study completion, an average of 6 months
Population: Safety population
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | RxSight RxLAL IOL
Number analyzed (Participants) | 51
Number analyzed (Eyes) | 101
Eyes | 3

3. Other Pre Specified Outcome: Number of Eyes That Received Secondary Surgical Interventions (SSIs)
Description: Secondary Surgical Interventions (SSIs) of the study eyes that occur during the conduct of the study.
Time Frame: Through study completion, an average of 6 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | RxSight RxLAL IOL
Number analyzed (Participants) | 51
Number analyzed (Eyes) | 101
Eyes | 1

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Description: Non-ocular, Non-serious adverse events were not required to be collected per protocol. All-Cause Mortality and Non-Ocular Serious Adverse Events are reported at the participants level. Ocular Serious and Other (Not Including Serious) Adverse Events are presented with total number of eyes monitored/assessed as the at Risk population.
Arm/Group | RxSight RxLAL IOL
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 2/101
Other Adverse Events (participants affected / at risk) | 28/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RxSight RxLAL IOL (N=101)
IOL Explant (Surgical and medical procedures) | 1 (1)
Gastritis with diarrhea (Gastrointestinal disorders) | 1/51 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RxSight RxLAL IOL (N=101)
Loss of BSCVA of ≥ 10 letters due to dry Eye (Eye disorders) | 2 (2) — Compared to postop week 3
Clinically significant cystoid macular edema (Eye disorders) | 2 (2)
Corneal Edema (Eye disorders) | 1 (1) — Corneal Edema (corneal swelling (stromal or epithelial) resulting in BCDVA ≤ 20/40 after Postop Week 3
Blurred vision right eye (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Cornea Epithelialized with SPK (Eye disorders) | 2 (2)
Diabetic macular edema (Eye disorders) | 3 (3)
Increased protein distribution after lock-in procedure (Eye disorders) | 1 (1)
Giant cells on anterior surface of IOL (Eye disorders) | 2 (2)
Non-clinically significant cystoid macular edema (Eye disorders) | 6 (6)
Posterior Capsular Opacity (Eye disorders) | 3 (3)
Loss of BCDVA due to Posterior Capsular Opacity (Eye disorders) | 2 (2) — Compared to postop week 3
Loss of BCDVA due to lens aberrations (Eye disorders) | 1 (1) — Compared to postop week 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: CSP-025-05 rev DE protocol and SAP 05-16-2019_Redacted (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03771352/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: CSP-025 rev 5 UK protocol and SAP 05-16-2019_Redacted (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03771352/Prot_SAP_001.pdf